CLINICAL TRIAL: NCT05206370
Title: A Second Multicenter, Double-blind, Randomized, Placebo-controlled Phase 3 Trial Evaluating the Efficacy and Safety of Cytisinicline in Adult Smokers
Brief Title: A Second Study of Cytisinicline for Smoking Cessation in Adult Smokers
Acronym: ORCA-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-CYT-04
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo + Behavioral Support (Placebo Comparator): One placebo tablet orally (PO) three times daily (TID) for 12 weeks plus behavioral support
  Interventions: Drug: Placebo; Behavioral: Behavioral support
- 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support (Experimental): One cytisinicline tablet PO TID for 6 weeks followed by one placebo tablet PO TID for 6 weeks plus behavioral support
  Interventions: Drug: Cytisinicline; Drug: Placebo; Behavioral: Behavioral support
- 12-Week Cytisinicline + Behavioral Support (Experimental): One cytisinicline tablet PO TID for 12 weeks plus behavioral support
  Interventions: Drug: Cytisinicline; Behavioral: Behavioral support

INTERVENTIONS:
Drug: Cytisinicline — film-coated oral tablets containing 3 mg cytisinicline
  Other Names: Cytisine
  Arms: 12-Week Cytisinicline + Behavioral Support; 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support
Drug: Placebo — film-coated oral tablets containing matched placebo
  Arms: 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support; Placebo + Behavioral Support
Behavioral: Behavioral support — Behavioral support sessions by a qualified study site staff member will be participant-driven and will include direct engagement with the subject about their attempt to quit smoking. Each session will last approximately 10 minutes.

SUMMARY:
This placebo-controlled Phase 3 study is being conducted at sites within the United States to evaluate 3 mg cytisinicline TID for treatment duration of 42 days/6 weeks and evaluate 3 mg cytisinicline TID for treatment duration of 84 days/12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age ≥ 18 years.
2. Current daily cigarette smokers (averaging at least 10 cigarettes per day upon completing a 7-day screening smoking diary) and who intend to quit smoking.
3. Expired air carbon monoxide (CO) ≥ 10 ppm.
4. Failed at least one previous attempt to stop smoking with or without therapeutic support.
5. Willing to initiate study treatment on the day after randomization and set a quit date within 5-7 days of starting treatment.
6. Willing to actively participate in the study's smoking cessation behavioral support provided throughout the study.
7. Able to fully understand all study requirements, willing to participate, and comply with dosing schedule.
8. Sign the Informed Consent Form.

Exclusion Criteria:

1. More than 1 study participant in same household during the 12-week treatment period.
2. Previous cytisinicline treatment in a prior clinical study or any other cytisine usage.
3. Known hypersensitivity to cytisinicline or any of the excipients.
4. Positive urinary drugs of abuse screen, determined within 28 days before the first dose of cytisinicline.
5. Clinically significant abnormal serum chemistry or hematology values within 28 days of randomization (ie, requiring treatment or monitoring).
6. Clinically significant abnormalities in 12-lead ECG determined after minimum of 5 minutes in supine position within 28 days of randomization (ie, requiring treatment or further assessment).
7. Recent history (within 3 months) of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident, or hospitalization for congestive heart failure.
8. Current uncontrolled hypertension (blood pressure ≥160/100 mmHg).
9. Currently psychotic or having had a psychotic event within 3 months. If any subject becomes psychotic during the study, they must be removed from treatment and/or additional study visits.
10. Currently having suicidal ideation or risk for suicide ("Yes" to either question 4 or question 5 OR "Yes" to any suicidal behavior question on the Columbia Suicide Severity Rating Scale [C-SSRS] with clear suicidal intent or previous attempt).
11. Current symptoms of moderate to severe depression (depression score ≥11on the HADS).
12. Renal impairment defined as a creatinine clearance (CrCl) <60 mL/min (estimated with the Cockroft-Gault equation).
13. Hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0 x the upper limit of normal (ULN).
14. Women who are pregnant or breast-feeding.
15. Male or female subjects of childbearing potential who do not agree to use acceptable methods of birth control during the study treatment period.
16. Participation in a clinical study with an investigational drug in the 4 weeks prior to randomization.
17. Treatment with other smoking cessation medications (bupropion, varenicline, nortriptyline, or any nicotine replacement therapy [NRT]) in the 4 weeks prior to randomization or planned use of these other smoking cessation medications during the study.
18. Use within the 2 weeks prior to randomization or planned use during the study of non-cigarette and/or noncombustible nicotine products (pipe tobacco, cigars, snuff, smokeless tobacco, hookah, e-cigarettes/vaping) or marijuana smoking or vaping.
19. Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cain, Vice-President Clinical Research, Study Director — Achieve Life Sciences, Inc.
Locations (12):
- United States (12):
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Affinity Health Corp, Oak Brook, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Global Medical Institutes LLC; Princeton Medical Institute, Princeton, New Jersey
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Intend Research, Norman, Oklahoma
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Health Research of Hampton Toads, Inc, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prochaska J, Rubinstein M, Perdok R, Blumenstein B, Jacobs C. Cytisinicline for smoking cessation in individuals with self-reported COPD: a post hoc analysis of the ORCA-2 and ORCA-3 trials. Thorax. 2026 Jan 15;81(2):164-169. doi: 10.1136/thorax-2025-223880. PMID 40962497
- [Derived] Rigotti NA, Benowitz NL, Prochaska JJ, Rubinstein M, Clarke A, Blumenstein B, Cain DF, Jacobs C. Cytisinicline for Smoking Cessation: The ORCA Phase 3 Replication Randomized Clinical Trial. JAMA Intern Med. 2025 Jun 1;185(6):648-655. doi: 10.1001/jamainternmed.2025.0628. PMID 40257755

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo + Behavioral Support | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support | 12-Week Cytisinicline + Behavioral Support
Started | 265 | 263 | 264
Completed | 209 | 207 | 212
Not Completed | 56 | 56 | 52
Not completed — Adverse Event | 3 | 4 | 5
Not completed — Withdrawal by Subject | 27 | 30 | 24
Not completed — Physician Decision | 1 | 3 | 2
Not completed — Death | 0 | 1 | 3
Not completed — Lost to Follow-up | 23 | 16 | 14
Not completed — Other, Nor Specified | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Behavioral Support: One placebo tablet PO TID for 12 weeks plus behavioral support
- Total: Total of all reporting groups
Arm/Group | Placebo + Behavioral Support | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support | 12-Week Cytisinicline + Behavioral Support | Total
Number analyzed (Participants) | 265 | 263 | 264 | 792
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11.4) | 52 (11.7) | 52 (12.3) | 52 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 142 | 151 | 439
  Male | 119 | 121 | 113 | 353
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 13 | 45
  Not Hispanic or Latino | 248 | 248 | 251 | 747
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 0 | 5
  Asian | 0 | 2 | 2 | 4
  Black or African American | 51 | 38 | 50 | 139
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  White | 210 | 216 | 205 | 631
  Other, Not Specified | 3 | 3 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Smoking Abstinence From Weeks 3 to Week 6
Description: Smoking abstinence as verified by weekly expired carbon monoxide (CO) measurements ≤ 10 parts per million (ppm).
Time Frame: Weeks 3 to 6
Population: All Randomized Set: all randomized participants. Placebo and 6-week treatment arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support
Number analyzed (Participants) | 265 | 263
percentage of participants | 6.0 | 14.8
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support; Test type: Superiority — Abstinence from Week 3 to Week 6; p = 0.0008, Exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 2.85, 95% CI 2-sided [1.475 to 5.617] — Common odds ratio (stratified by site)
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support; Test type: Superiority; p = 0.0010, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.485 to 5.094] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel — p-value for difference in proportions; Difference in proportions = 0.09, 95% CI 2-sided [0.033 to 0.134]

2. Primary Outcome: Percentage of Participants With Smoking Abstinence From Weeks 9 to Week 12
Description: Smoking abstinence as verified by weekly expired CO measurements ≤ 10 ppm.
Time Frame: Weeks 9 to 12
Population: All Randomized Set: all randomized participants, Placebo and 12-week treatment arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | 12-Week Cytisinicline + Behavioral Support
Number analyzed (Participants) | 265 | 264
percentage of participants | 9.4 | 30.3
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs 12-Week Cytisinicline + Behavioral Support; Abstinence from Week 9 to Week 12; Test type: Superiority; p < 0.0001, Exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 4.40, 95% CI 2-sided [2.566 to 7.343] — Common odds ratio (stratified by site)
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs 12-Week Cytisinicline + Behavioral Support; Test type: Superiority; p < 0.0001, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 4.17, 95% CI 2-sided [2.575 to 6.885] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs 12-Week Cytisinicline + Behavioral Support; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — p-value for difference in proportions4; Difference in proportions = 0.21, 95% CI 2-sided [0.141 to 0.267]

3. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 3 to Week 24
Description: Smoking abstinence as verified by expired CO measurements ≤ 10 ppm. Measurements were weekly from Week 3 to Week 12 and monthly from Week 12 to Week 24.
Time Frame: Week 3 to Week 24
Population: All Randomized Set: all randomized participants, Placebo and 6-week treatment arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support
Number analyzed (Participants) | 265 | 263
percentage of participants | 1.1 | 6.8
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support; Abstinence from Week 6 to Week 24; Test type: Superiority; p = 0.0006, Exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 6.25, 95% CI 2-sided [1.851 to 34.619] — Common odds ratio (Stratified by site)
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support; Test type: Superiority; p = 0.0007, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 6.42, 95% CI 2-sided [2.026 to 27.544] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel — p-value for difference in proportions; Difference in proportions = 0.06, 95% CI 2-sided [0.023 to 0.075]

4. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 9 to Week 24
Description: Smoking abstinence as verified by expired CO measurements ≤ 10 ppm. Measurements were weekly from Week 9 to Week 12 and monthly from Week 12 to Week 24.
Time Frame: Week 9 to Week 24
Population: All Randomized Set: all randomized participants, Placebo and 12-week treatment arms only.
Measure: Number; unit: percentage of participants
Groups:
- Cytisinicline + Behavioral Support: One cytisinicline tablet PO TID for 12 weeks plus behavioral support
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Number analyzed (Participants) | 265 | 264
percentage of participants | 4.2 | 20.5
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Abstinence from Week 9 to Week 24; Test type: Superiority; p < 0.0001, Exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 5.79, 95% CI 2-sided [2.888 to 12.458] — Common odds ratio (stratified by site)
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Test type: Superiority; p < 0.0001, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 5.94, 95% CI 2-sided [3.091 to 12.130] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — p-value for difference in proportions; Difference in proportions = 0.16, 95% CI 2-sided [0.110 to 0.202]

5. Secondary Outcome: Percentage of Participants Taking Cytisinicline Who Are Relapse-Free at Week 24
Description: Relapse is defined as participant reported resuming smoking or an expired CO measure ≥ 10 ppm. Relapse is defined as a participant having met one of the following: not being abstinent from Weeks 3 to 6; not being abstinent at the Week 12 visit; not being abstinent or not self-reporting abstinence during the Week 16 to Week 24 follow-up period. (During the follow-up period [Weeks 16 to 24], up to a total of 5 cigarettes could have been smoked.)
Time Frame: Week 24
Population: All Randomized Set: All randomized participants. Participants in the cytisinicline arms.
Measure: Number; unit: percentage of participants
Arm/Group | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support | 12-Week Cytisinicline + Behavioral Support
Number analyzed (Participants) | 263 | 264
percentage of participants | 8.7 | 10.6
Statistical Analysis 1: Comparison: 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support vs 12-Week Cytisinicline + Behavioral Support; Relapse free at Week 24; Test type: Superiority; p = 0.5538, Exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.652 to 2.297] — Common odds ratio (stratified by site)
Statistical Analysis 2: Comparison: 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support vs 12-Week Cytisinicline + Behavioral Support; Test type: Superiority; p = 0.5560, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.691 to 2.231] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support vs 12-Week Cytisinicline + Behavioral Support; Test type: Superiority; p = 0.2822, Zelen's exact test (Pr ≤ P)

ADVERSE EVENTS:
Time Frame: From signing of informed consent through Week 24
Description: Safety Set: participants who received study drug
Arm/Group | Placebo + Behavioral Support | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support | 12-Week Cytisinicline + Behavioral Support
All-Cause Mortality (participants affected / at risk) | 0/262 | 1/263 | 3/260
Serious Adverse Events (participants affected / at risk) | 8/262 | 8/263 | 8/260
Other Adverse Events (participants affected / at risk) | 110/262 | 132/263 | 137/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Behavioral Support (N=262) | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support (N=263) | 12-Week Cytisinicline + Behavioral Support (N=260)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Hernia (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Per investigator assessment, resulting death was considered unrelated or unlikely to be associated with cytisinicline treatment.
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Per investigator assessment, resulting death was considered unrelated or unlikely to be associated with cytisinicline treatment.
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Per investigator assessment, resulting death was considered unrelated or unlikely to be associated with cytisinicline treatment.
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 — Per investigator assessment, resulting death was considered unrelated or unlikely to be associated with cytisinicline treatment.
Migraine with aura (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Behavioral Support (N=262) | 6-Week Cytisinicline + 6-Week Placebo + Behavioral Support (N=263) | 12-Week Cytisinicline + Behavioral Support (N=260)
Constipation (Gastrointestinal disorders) | 3 | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 12 | 12 | 8
Dry mouth (Gastrointestinal disorders) | 6 | 12 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 6 | 5
Nausea (Gastrointestinal disorders) | 19 | 26 | 19
Vomiting (Gastrointestinal disorders) | 6 | 2 | 3
Fatigue (General disorders) | 3 | 7 | 11
Bronchitis (Infections and infestations) | 7 | 2 | 2
COVID-19 (Infections and infestations) | 27 | 18 | 27
Gastroenteritis viral (Infections and infestations) | 3 | 0 | 7
Nasopharyngitis (Infections and infestations) | 7 | 2 | 3
Sinusitis (Infections and infestations) | 6 | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 11 | 12
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2 | 1
Increased appetite (Metabolism and nutrition disorders) | 3 | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 10 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 6
Dizziness (Nervous system disorders) | 2 | 3 | 10
Headache (Nervous system disorders) | 18 | 21 | 22
Abnormal dreams (Psychiatric disorders) | 16 | 24 | 20
Anxiety (Psychiatric disorders) | 6 | 8 | 6
Depression (Psychiatric disorders) | 6 | 6 | 5
Insomnia (Psychiatric disorders) | 20 | 29 | 32
Irritability (Psychiatric disorders) | 3 | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 2
Hypertension (Vascular disorders) | 13 | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT05206370/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT05206370/SAP_001.pdf